CLINICAL TRIAL: NCT04013737
Title: Enhanced, Personalized and Integrated Care for Infection Management at the Point-Of-Care
Acronym: EPICIMPOC
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 16HH3526
Record Dates: First submitted 2019-01-31; First posted 2019-07-10 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Antibiotic Resistant Infection; Infection
Keywords: Antimicrobial Resistance; Antibiotic prescribing; Clinical Decision Support Systems
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients and Public: Exploration of patient and public engagement with antibiotic decision making in secondary care. Prospective evaluation of a co-designed intervention to support enhanced knowledge and understanding of infections and their management.
  Interventions: Device: EPIC IMPOC
- Prescribers: Quantitative evaluation of the impact of using a clinical decision support system to support antibiotic decision making.
  Interventions: Device: EPIC IMPOC

INTERVENTIONS:
Device: EPIC IMPOC — Clinical Decision Support System for antibiotic prescribing.

SUMMARY:
Antimicrobials (drugs that kill or stop the growth of microorganisms including bacteria, thereby treating infections) commonly used to treat patients with infections are becoming less effective over time as bacteria develop resistance to them. Antimicrobial usage itself can lead to development and spread of antimicrobial resistance. Antimicrobial resistance is now a major threat to patient safety. To conserve the effectiveness of antimicrobials the investigator need to develop ways to use them more sensibly healthcare professionals who diagnose and treat infections must be able to access antimicrobial guidelines and test results at the patient bedside. This needs to be provided rapidly and with support to make sure that the decisions on prescribing antimicrobials are the best that can be made.

DETAILED DESCRIPTION:
Prototype software to achieve this has been developed through collaboration between healthcare professionals and biomedical engineers. This prototype software (run on a mobile device) retrieves patient results from various laboratory and clinical databases (securely within the Trust firewall) and displays this to the clinician making the prescribing decision. Furthermore a machine learning algorithm is applied to the data, and similar anonymised historical cases (and the antimicrobials prescribed and the clinical outcomes) are also displayed to the clinician to further inform their decision making. The prototype has been designed for use in intensive care, where the risk of infection is high, but through the research project detailed here, the software will be developed and validated across other areas of hospital patient care. Furthermore there is a key need to engage patients with how decisions are made around antimicrobial prescribing. The investigator propose to adapt the prototype to meet these needs. This system should improve patient safety and help preserve the effectiveness of existing antimicrobials

ELIGIBILITY:
Inclusion Criteria:

(i) healthcare professionals for evaluation phases: Have read the PIL and consent to participate in the study

(ii) patients for whom the clinician chooses to use the POC DSS as a resource when prescribing antimicrobials: Adult patients > 18 years old Being managed for infection outside of the critical care setting in Imperial College Healthcare NHS Trust Deemed appropriate for management with POC DSS by attending physician Prescribed antimicrobial agents outside of the critical care setting in last 5 days

(iii) Prescriber / healthcare professional for using POC DSS: Trained Healthcare Professional Working within wards under assessment Deemed suitable for recruitment by senior member of their team

Exclusion Criteria:

(i) healthcare professionals: Do not wish to participate in the study Working across wards which is acting as a control ward Deemed no suitable for recruitment by a senior member of their team Non-permanent member of the Trust Information governance training not up-to-date

(ii) patients recruits Critical care patients Paediatric patients < 18 years old Deemed not suitable for management using POC DSS by attending physician On palliative care, end of life pathway Prisoners / young offenders in custody of HM Prison Service Involved in current research or have recently been involved in any research prior to recruitment (last 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients may be asked to participate in the evaluation of the the patient module.
  For prescriber recruitment to use the application the following methods of identifying participants will be undertaken:
  Phase 1: Participants will be identified based on their roles within the infectious disease team (level and areas of the hospital covered) and will be directly approached by the study PI / clinical infection lead to request their support with this phase of the project.
  Phase 2: Participants (physicians) will be identified based on the wards that they work in.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Holmes, Principal Investigator — Professor
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be considered on individual request in accordance with local information governance and research ethics approvals.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Professionals recruited = 15 Patients recruited for prospective study of engagement tool = 18
Pre-assignment Details: 15 healthcare professionals were recruited who would be using the tool to make antibiotic prescribing decisions.
  18 patients were enrolled in the pre- post- assessment of the impact of a patient-communication tool within the system on knowledge and understanding of their infection and its management.
Groups:
- Patients and Public: Prospective evaluation of knowledge and understanding of infections pre- and post- a patient communication intervention.
Period: Overall Study
Arm/Group | Patients and Public | Prescribers
Started | 18 | 15
Completed | 18 (12 participants declined to participate in the study) | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants that consented to participate
Groups:
- Patients and Public: Exploration of patient and public engagement with antibiotic decision making in secondary care. Qualitative evaluation and co-design of interventions. Prospective evaluation of intervention.
  EPIC IMPOC: Clinical Decision Support System for antibiotic prescribing.
- Prescribers: Quantitative and qualitative evaluation of the impact of using a clinical decision support system to support antibiotic decision making.
  EPIC IMPOC: Clinical Decision Support System for antibiotic prescribing.
- Total: Total of all reporting groups
Arm/Group | Patients and Public | Prescribers | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Median (Full Range); unit: Years] — Population: Age not collect
  Years
    number analyzed (Participants) | 18 | 0 | 18
    (all) | 66 [22 to 85] |  | 66 [22 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 10 | 8 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Appropriate Antimicrobial Prescriptions Recommended
Description: This will be measured by assessing the appropriateness of prescriptions recommended by the system compared to current clinical practice. Appropriateness is determined by evaluating prescribing against current clinical guidelines or infection expert opinion on best practice and is expressed as a proportion of the total number of antibiotic prescriptions made. Each individual patient has a single antibiotic prescription evaluated.
Time Frame: Single prescription at the time of antimicrobial prescribing assessment (e.g. at the time antibiotics were prescribed)
Population: 15 prescribers made 224 antimicrobial prescriptions during the study period which were analysed for the outcome measure.
Measure: Number; unit: percentage of prescriptions appropriate
Units Other Than Participants: Prescriptions made by participants
Groups:
- Appropriateness of Antibiotic Prescribing: Proportion of appropriate recommendations made using the case-based-reasoning algorithm out of 224 prescriptions input into the system by participants.
Arm/Group | Appropriateness of Antibiotic Prescribing
Number analyzed (Participants) | 15
Number analyzed (Prescriptions made by participants) | 224
percentage of prescriptions appropriate | 90

2. Primary Outcome: Evaluation of Effectiveness Assessed by User Acceptance of the Device
Description: This was assessment was a single time point at baseline (Pre-intervention) and single time point after use of the device in the study.
  Scores were pre-determined based on anticipated answers provided by participants pre- and post- intervention using a bespoke mark scheme (https://aricjournal.biomedcentral.com/articles/10.1186/s13756-018-0333-1).
  Participants could score between 0 (lowest) and 13 (highest) marks based on their responses to questions assessing knowledge and understanding.
Time Frame: Single time point before and after use of the device in the study
Population: Patients in hospital.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Improvement in Short Term Knowledge/Understanding: Compared using pre- and post- intervention questionnaire
Arm/Group | Improvement in Short Term Knowledge/Understanding
Number analyzed (Participants) | 18
score on a scale
  Pre-intervention | 3 [2 to 5]
  Post-intervention | 10 [6 to 11]

ADVERSE EVENTS:
Time Frame: Not assessed
Description: Adverse events were not assessed as this was not an observational study.
Arm/Group | EG000
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04013737/Prot_SAP_000.pdf